CLINICAL TRIAL: NCT01096082
Title: Randomized Clinical Trial to Assess the Safety and Efficacy of Lithium Carbonate in Patients With Spinocerebellar Ataxia Type 3
Brief Title: Safety and Efficacy of Lithium Carbonate in Patients With Spinocerebellar Ataxia Type 3
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Principal Investigator, Laura Bannach Jardim, MD PhD, Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09-418; HCPA FIPE GPPG: 09-418 (Other Grant/Funding Number: HCPA FIPE GPPG: 09-418)
Record Dates: First submitted 2010-03-29; First posted 2010-03-30 (Estimated); Last update posted 2013-01-30 (Estimated); Status verified 2013-01

CONDITIONS: Spinocerebellar Ataxia Type 3; Machado Joseph Disease
Keywords: spinocerebellar ataxia; Treatment; Lithium carbonate
MeSH Terms: conditions — Machado-Joseph Disease; Spinocerebellar Ataxias | interventions — Lithium Carbonate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Lithium Carbonate (Experimental)
  Interventions: Drug: Lithium Carbonate

INTERVENTIONS:
Drug: Lithium Carbonate — 300 mg tablets, starting dose 300 mg/day
  Arms: Lithium Carbonate
Drug: Placebo — Similar shape, color and taste and the same number of tablets from the experimental group
  Arms: Placebo

SUMMARY:
Design: Phase II-III, double-blind, parallel, placebo controlled randomized Clinical trial

Background: Spinocerebellar ataxia type 3 (SCA-3) is an autosomal dominant adult-onset neurodegenerative disorder for which there is no current treatment. Patients will invariably become dependent from others and unable to walk during the disease course.

Hypothesis: Lithium Carbonate is safe and effective in treating neurological symptoms and improving quality of life of patients with SCA3.

Outcomes:

Primary

* Phase 2 - To assess safety and tolerability of Lithium Carbonate in patients with SCA3 after 6 months of follow-up
* Phase 3 (if Phase II study shows safety of therapy) - To assess efficacy of Lithium Carbonate in patients with SCA3 through the Neurological Examination Score for SCA 3 (NESSCA) after 12 months of follow-up .

Secondary

1. - To assess efficacy on neurological function, ataxic, depressive and quality of life scores of Lithium Carbonate in patients with SCA3 through the Scale for the Assessment and Rating of Ataxia (SARA), 9-Hole Peg Board test, 8m walking time, PATA repetition rate, Click Test, SCA Functional Index (SCAFI), Composite Cerebellar Functional Score (CCFS), Beck Depression Inventory, Barthel Index and WHOQol after 6 and 12 months of follow-up.
2. - To assess the effect of Lithium Carbonate in peripheral levels and expression of treatment biomarkers (BDNF, NSE, HDAC, GSK-3Beta)

Study Duration: 12 months

* Final analysis of phase 2 (safety study) at 6 months with continuous monitoring until the end of phase 3 (efficacy study).
* Preliminary analysis of efficacy on ataxia scales at 6 months of study and final analysis of phase 3 at 12 months.

Obs: A futility analysis will be performed after 12 months of therapy if no statistically significant difference between groups were found. This analysis will define if the study will continue until 18 or 24 months of follow-up or will be ended at 12 months.

Location: Hospital de Clínicas de Porto Alegre

Subjects: 60 molecularly diagnosed SCA3 patients from the outpatient unit of the Medical Genetics Service of Hospital de Clínicas de Porto Alegre

Intervention: Lithium Carbonate tablets of 300mg. Starting dose will be 300mg/day with drug titration during 49 days or until achieving the defined target lithium serum level of 0.5 to 0.8 mEq/L

ELIGIBILITY:
Inclusion Criteria:

* Prior molecular diagnose of SCA3 with determined number of CAG expanded repeat.
* Not restricted to wheelchair.
* With disease duration between 2 and 10 years and more than 16 years old.

Exclusion Criteria:

* Signs of cardiopathy, elevated levels of creatinine, transaminases, bilirubins more than 1.5 times the normal upper limit at baseline.
* History of previous lithium carbonate significant adverse reaction, or drug abuse or alcoholism.
* Disturbance of thyroid function at baseline.
* Participation on another clinical trial less than 4 weeks before the study entrance.
* Current use of valproic acid, memantine, neuroleptics and anticoagulants
* If the individual (woman) did not agree in utilize a high effective contraceptive method during the study period and 3 months after the study-end.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2011-05; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Phase 2 - Safety and tolerability of Lithium Carbonate treatment in patients with SCA3 | 6 months
  According to the Common toxicity criteria manual, version 2.0
Phase 3 - Efficacy of Lithium Carbonate treatment in patients with SCA3 | 12 months
  Application of the Neurological Examination Score for SCA 3 (NESSCA)

SECONDARY OUTCOMES:
Efficacy of Lithium Carbonate in patients with SCA3 on neurological function, ataxic, depressive and quality of life scores | 6 and 12 months
  Scale for the Assessment and Rating of Ataxia (SARA), 9-Hole Peg Board test, 8m walking time, PATA repetition rate, Click Test, SCA Functional Index (SCAFI), Composite Cerebellar Functional Score (CCFS), Beck Depression Inventory, Barthel Index and WHOQol
Effect of Lithium Carbonate treatment in peripheral levels and expression of treatment biomarkers | 3 and 6 months
  BDNF, NSE, HDAC, GSK-3Beta

CONTACTS AND LOCATIONS:
Overall Officials: Laura B Jardim, MD PhD, Principal Investigator — Medical Genetics Service Hospital de Clinicas de Porto Alegre; Jonas AM Saute, MD, Study Director — Neurology Service Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Background] Watase K, Gatchel JR, Sun Y, Emamian E, Atkinson R, Richman R, Mizusawa H, Orr HT, Shaw C, Zoghbi HY. Lithium therapy improves neurological function and hippocampal dendritic arborization in a spinocerebellar ataxia type 1 mouse model. PLoS Med. 2007 May;4(5):e182. doi: 10.1371/journal.pmed.0040182. PMID 17535104
- [Derived] Saute JA, Rieder CR, Castilhos RM, Monte TL, Schumacher-Schuh AF, Donis KC, D'Avila R, Souza GN, Russo AD, Furtado GV, Gheno TC, Souza DO, Saraiva-Pereira ML, Portela LV, Camey S, Torman VB, Jardim LB. Planning future clinical trials in Machado Joseph disease: Lessons from a phase 2 trial. J Neurol Sci. 2015 Nov 15;358(1-2):72-6. doi: 10.1016/j.jns.2015.08.019. Epub 2015 Aug 14. PMID 26297649
- [Derived] Saute JA, de Castilhos RM, Monte TL, Schumacher-Schuh AF, Donis KC, D'Avila R, Souza GN, Russo AD, Furtado GV, Gheno TC, de Souza DO, Portela LV, Saraiva-Pereira ML, Camey SA, Torman VB, de Mello Rieder CR, Jardim LB. A randomized, phase 2 clinical trial of lithium carbonate in Machado-Joseph disease. Mov Disord. 2014 Apr;29(4):568-73. doi: 10.1002/mds.25803. Epub 2014 Jan 7. PMID 24399647